CLINICAL TRIAL: NCT06870136
Title: A Direct-to-Consumer, Randomized, Double-blind, Placebo-controlled Study Evaluating the Quality and Effects of Lion's Mane Product on Cognitive Health Outcomes Through Self-Reported Measures
Brief Title: Study Evaluating the Quality and Effects of Lion's Mane Product on Cognitive Health
Status: Recruiting | Type: Observational
Sponsor: M2 Ingredients (Industry)
Responsible Party: Sponsor
Other Study IDs: PS14
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lion's Mane Study Product: Participants will be randomized to one of two groups A or B: (1) Lion's Mane Study Product, and (2) Placebo. The Investigators and study team and participants will be blinded to the group assignment.
  Interventions: Dietary Supplement: Lion's Mane Study Product
- Placebo: Participants will be randomized to one of two groups A or B: (1) Lion's Mane Study Product, and (2) Placebo. The Investigators and study team and participants will be blinded to the group assignment.

INTERVENTIONS:
Dietary Supplement: Lion's Mane Study Product — The Lion's Mane Study product contains vegetable cellulose (capsules), Certified organic Lion's Mane (Hericium erinaceus) fruiting body and mycelial biomass cultured on certified whole oats (Avena sativa). Screening assessments, scales and surveys during baseline and during the use of the study product/placebo and end of study experience survey data will be collected.
  Groups: Lion's Mane Study Product

SUMMARY:
The rationale for this study is to observe differences in cognitive health outcomes such as short term memory and simple reaction time between a consumer-grade and commercially available Lion's mane mushroom product and a placebo control group. Additionally, the study aims to evaluate the impact of the product on cognitive function, mood, focus, motivation, sleep quality, and stress. A consumer-driven, decentralized observational clinical research study is therefore well-suited for evaluating the impact of this product in this population.

The study will evaluate cognitive health outcomes in a broad age-range of adults who have chosen to try this product. The study will incorporate memory and cognitive function tests, participant reported outcome questionnaires and surveys. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and participate in the observational process with self-reported measures that can be done at home. Findings from this study will contribute knowledge toward the functional mushrooms and cognitive health and the design of future studies.

DETAILED DESCRIPTION:
Mushrooms from the genera Hericium are among the many mushrooms known for their long history of traditional use. Hericium erinaceus (commonly known as Lion's Mane) is a wood-decaying basidiomycete that can grow on many tree species including birch, oak, maple, and beech trees. The fruiting body is white when fresh and yellowish with age. It consists of a rounded solid mass of spines that are 1-4cm long which hang down in a beardlike fashion. The mushroom is attached to the tree by a tough, thick, root-like structure.

H. erinaceus has been reported to have immunomodulatory, neurotrophic, neuroprotective, antioxidant, anti-tumor, anti-inflammatory, prebiotic, and gut-health promoting effects. The principal components of medical interest include polysaccharides, glycoproteins, hericenones, erinacines, and hericerin.

Previous work has shown mood-enhancing effects following chronic administration of H.

erinaceus with both studies showing improvements in depression and anxiety scores. More recently, a study on the acute and chronic effect of H. erinaceus suggested that it may improve speed of performance and reduce subjective stress in healthy, young adults. Similarly, another recent study observed improvements in cognitive function and changes in circulating brain-derived neurotrophic factor (BDNF) levels supporting the proposed neurotrophic and neuroprotective effects of the bioactive metabolites present in H. erinaceus. When looking specifically at the impact of H. erinaceus on memory, another study showed that oral intake of H. erinaceus significantly improved cognitive functions and prevented the deterioration of memory over time. Given the previous work in the literature on older adults and adults with comorbidities, there is a need to understand the benefits of H. erinaceus on cognitive health in a healthy adult population. In addition, given the variety of products on the market and the unique fingerprint of bioactive molecules in the mycelium and the fruit body of H. erinaceus, a study where the treatment consisted on both the mycelium and the fruit body would be beneficial to understanding this popular nutraceutical ingredient.

H. erinaceus is a popular culinary mushroom species that is wild-harvested and cultivated in many countries. Thus, preparations made from liquid fermentation or solid-state fermentation processes provides a means to highly efficient, consistent, year-round production and allow for better quality control of the final product. The preparation used in this study is a certified organic powdered H. erinaceus (Strain M2-102-10) mycelial biomass and fruiting body cultured on organic whole oats (Avena sativa) in a controlled solid fermentation facility. The powder was encapsulated in vegetable cellulose capsules and each dose consisted of 2g of powder (3 capsules).

ELIGIBILITY:
Inclusion Criteria:

* Individuals 40-75 years old, inclusive
* Has self-reported concerns with reduced memory, focus and cognitive decline
* Cognitive Failures Questionnaire score of mild to moderate at screening
* Interested in understanding more about their cognitive health and have chosen have chosen to use the study product
* Willing to do a 4-week washout from any supplements for memory or cognitive function prior to randomization
* Willing to do a 4-week washout prior to randomization from supplements with mushroom compounds or consuming mushrooms known to impact NGF. This includes but may not be limited to: Reishi (ganoderma lucidum), cordyceps (cordyceps militaris or cordyceps sinensis), Lion's mane or Coral Tooth Fungus (hericium coralloides), turkey tail (trametes versicolor), Chage (inonotus obliquus), Maitake (grifola frondosa).
* If taking prescription medications for sleep (e.g. Benzodiazepines, zolpidem, zaleplon), or other class of medication for sleep, must be on a "stable dose" for at least 4 weeks prior to enrollment. "Stable dose" is defined as no changes in dosage or frequency of the specified medications for at least 4 weeks prior to enrollment and throughout the study period.
* If regularly consuming alcohol, must be willing to stay on a stable amount throughout the study period and to log alcohol consumption.
* In good general health at the time of screening (Investigator discretion).
* Able to read and understand English.
* Able to read, understand, and provide informed consent.
* Able to use a personal smartphone device and laptop, download Chloe by People Science and use the BrainHQ web-based assessment platform.
* Able to receive shipment of the product at an address within the United States.
* Able to complete study assessments over the course of up to 9 weeks.

Exclusion Criteria:

Any potential participants who:

* Do not have a smartphone and/or internet access.
* Concomitant Therapies:

  * Participants taking prescription medication for sleep (e.g. Benzodiazepines, zolpidem, zaleplon) not on a stable dose for at least 4 weeks
  * Participants receiving Cognitive Behavioral Therapy for Insomnia (CBTi)
  * Participants receiving any investigational therapies or treatments within 30 days prior to randomization.
* Other Illnesses or Conditions: Participants who have the following conditions or comorbidities are excluded:

  * Diagnosis of Alzheimer's disease or dementia
  * Diagnosed neurological condition or assessed as having a learning/behavioural or neurodevelopmental difference such as dyslexia or ADHD
  * Have a visual impairment that cannot be corrected with glasses or contact lenses, including red green color blindness
  * Deafness or untreated age-related hearing loss
  * Confirmed diagnoses of the following sleep disorders: Narcolepsy, Restless Leg Syndrome, Circadian Rhythm Disorders
  * Current or prior history of psychotic disorder
  * Diagnosed with Alcohol or Substance Abuse Disorder
  * Currently pregnant, planning to become pregnant at any time during the study, or breastfeeding
  * Have a significant illness, disease or condition which, in the opinion of the principal investigator, may impact their ability to participate in the trial or impact the trial outcomes
  * Long Covid including persistent feelings of brain fog
  * Participants using any nicotine and cannabis-containing products
  * Known hypersensitivity or previous allergic reaction to Lion's mane or functional mushrooms.
  * Are unlikely for any reason to be able to comply with the trial or considered unsuited for participation in the study by the Principal Investigator.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants between 40-75 years old experiencing reduced memory, focus, and cognitive decline. Participants will be recruited through People Science community, email outreach, physician network, advocacy groups and social media channels. Advertisements will be in digital format and will link to a study landing page to enable participant sign-up where they will complete a pre-screening qualification survey.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Impact on Attention, Short Term & Working Memory | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The primary outcome measure is to evaluate the impact of the Lion's Mane study product on a composite measure of Attention, Short Term & Working Memory. This will be measured using the change from baseline in BrainHQ Cognitive Test Suite composite score at Week 8 between placebo and study product group.

SECONDARY OUTCOMES:
Fluid intelligence and spatial memory | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary outcome will be to evaluate the impact of the Lion's mane study product on fluid intelligence and spatial memory. This will be measured using the change in overall fluid intelligence and spatial memory between placebo and study product group between placebo as measured by Sandia's progressive matrices, spatial memory and visual search task, grid memory task and shape rotation score. Baseline period will be compared as well.
Multiple object tracking, Visual and Numerical tasks | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary outcome will be to evaluate the impact of the Lion's mane study product on multiple object tracking, visual and numerical tasks. This will be done using the change in cognitive function as measured by Cognitive Failures Questionnaire score between placebo and study product group. Baseline period will be compared as well.
Subjective awareness of cognitive failures | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary outcome will be to evaluate the impact of the Lion's mane study product on subjective awareness of cognitive failures. This will be done using the change in average mood score as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Mood perception | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary outcome will be to evaluate the impact of the Lion's mane study product on mood perception. This will be done using the change in average subjective focus as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Perception of focus | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary outcome will be to evaluate the impact of the Lion's mane study product on perception of focus. This will be done using the change in average subjective motivation as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Subjective Motivation | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary objective will be to evaluate the impact of the Lion's mane study product on subjective motivation. This will be done using the change in average subjective motivation as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Sleep quality | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary objective will be to evaluate the impact of the Lion's mane study product on sleep quality. This will be done using the change in average sleep quality score as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Daytime alertness | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary objective will be to evaluate the impact of the Lion's mane study product on daytime alertness. This will be done using the change in average daytime alertness score as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.
Stress | Participants will complete up to a 14-week study consisting of screening period, randomization and shipping period, a baseline period, and an 8-week product/placebo use period.
  The secondary objective will be to evaluate the impact of the Lion's mane study product on stress. This will be done using the change in average stress score as measured by a daily 10-point visual analogue rating scale (VAS) between the study product and placebo group Baseline period will be compared as well.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Kazaryan, MPhil, Study Director — People Science, Inc.
Locations (1):
- People Science, Los Angeles, California, United States